CLINICAL TRIAL: NCT05589337
Title: Effects of Baduanjin Breathing Training for Depression and Anxiety Patients: a Prospective Randomized Study
Brief Title: Baduanjin Training for Depression and Anxiety Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Lu Ying, MM, Research Associate, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202040253
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Depression Symptoms; Anxiety Symptoms
Keywords: Baduanjin; Depression; Anxiety; Randomized controlled trial
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a 16-week, randomized controlled trial. Patients with depression and anxiety symptoms are randomized to either Baduanjin intervention group or health education control group.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors were blinded to the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin intervention group (Experimental): Participants randomized to Baduanjin intervention group receive health education plus a Baduanjin training program. The Baduanjin training program was a 16-week, instructor-led group training program that offers breathing training as a core skill.
  Interventions: Behavioral: Baduanjin; Behavioral: Health education
- Health education control group (Active Comparator): Participants randomized to the health education control group only receive health education and no additional training program.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Baduanjin — The Baduanjin training program consisted of two 90-min training classes and at least five 30-min at-home practice sessions per week for 16-weeks. All sessions included 10 min of warmup and 10 min of cooldown.
  Other Names: Eight-section Brocade
  Arms: Baduanjin intervention group
Behavioral: Health education — Health education is provided by psychologist and TCM doctor, including work, rest, diet and other basic programs.

SUMMARY:
In recent years, the number of people with symptoms of depression or anxiety are on the rise. The aims of the prospective randomized study are: (1) to examine the effects of Baduanjin breathing training on reducing symptoms of depression or anxiety, and (2) to explore the correlates between improvements of depression or anxiety symptom and changes of lung functions.

DETAILED DESCRIPTION:
Depression and anxiety, the two common mental health problems, are prevalent in the world. But there is a lack of sufficient no-drug intervention for relieving these two symptoms. The study focuses on mixed depressive and anxiety disorder, which symptoms are not sufficiently severe, numerous, or persistent to justify a diagnosis of depressive disorder or an anxiety disorder.

Baduanjin is a form of mind-body exercise with a profound philosophical foundation rooted in oriental culture. Previous studies have provided some evidences of beneficial effects on Baduanjin for depression and anxiety. Moreover, the effects and mechanisms of Baduanjin on patients with symptoms of depression and anxiety are yet to be further investigated.

This is a two-group prospective, randomized, assessor-blinded trial, planning to enroll 120 participants (60 for Baduanjin intervention group receiving health education plus a Baduanjin breathing training program, and 60 for health education control group only receiving health education).

The aims of the prospective randomized study are: (1) to examine the effects of Baduanjin breathing training on reducing symptoms of depression or anxiety, and (2) to explore the correlates between improvements of depression or anxiety symptom and changes of lung function.

ELIGIBILITY:
Inclusion Criteria:

* Subject with depression or anxiety symptom diagnosed by ICD-10.
* Depression 7≤HAMD-17≤29，anxiety 7≤HAMA-14≤29.
* Subject has a clear mind and the ability to read, to talk and to communicate.
* Subject agrees to participate in this study and sign to the informed consent.

Exclusion Criteria:

* Subject with bipolar disorder, psychotic disorder, organic mental disorder and cognitive disorder.
* Subject with alcohol abuse, substance dependence and suicidal behavior in past-year.
* Subject has severe somatic disease.
* Subject is pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale | Change from Baseline HAMD-17 at 16 weeks
  The HAMD-17 is a clinician-rated assessment (structured interview) of patients' depressive symptoms. Questions focus on depressive symptoms during the past 7 days, and higher cumulative scores indicate more severe depression.
14-item Hamilton Anxiety Rating Scale | Change from Baseline HAMA-14 at 16 weeks
  The HAMA-14 is a clinician-rated assessment (structured interview) of patients' anxious symptoms. Questions focus on anxious symptoms during the past 7 days, and higher cumulative scores indicate more severe anxiety.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale-21 item | Change from Baseline DASS-21 at 8 weeks
  The DASS-21 is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Depression, Anxiety and Stress Scale-21 item | Change from 8 weeks DASS-21 at 16 weeks
  The DASS-21 is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Vital capacity | Change from Baseline VC at 16 weeks
  Vital capacity (VC) is tested by spirometry in the same machine (MINATO AS-507, Japan) and by the same clinicians following a standard protocol.
Forced vital capacity | Change from Baseline FVC at 16 weeks
  Forced vital capacity (FVC) is tested by spirometry in the same machine (MINATO AS-507, Japan) and by the same clinicians following a standard protocol.
FVC percentage of predicted normal values | Change from Baseline FVC% at 16 weeks
  FVC percentage of predicted normal values (FVC%) is tested by spirometry in the same machine (MINATO AS-507, Japan) and by the same clinicians following a standard protocol.
Forced expiratory volume in one second | Change from Baseline FEV1 at 16 weeks
  Forced expiratory volume in one second (FEV1) is tested by spirometry in the same machine (MINATO AS-507, Japan) and by the same clinicians following a standard protocol.
The ratio of FEV1 to FVC | Change from Baseline FEV1/FVC at 16 weeks
  The ratio of FEV1 to FVC (FEV1/FVC) is tested by spirometry in the same machine (MINATO AS-507, Japan) and by the same clinicians following a standard protocol.
Respiration rates | Change from Baseline respiration rates at 16 weeks
  The respiration rates are recorded by the same equipment (BioHarness, USA) and by the same clinicians following a standard protocol.
Respiration depths | Change from Baseline respiration depths at 16 weeks
  The respiration depths are recorded by the same equipment (BioHarness, USA) and by the same clinicians following a standard protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoting Zhao, Study Chair — Shanghai Qigong Research Institute; Ying Lu, Principal Investigator — Shanghai Qigong Research Institute; Jie Li, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai Qigong Research Institute, Shanghai, Shanghai Municipality, China